CLINICAL TRIAL: NCT07043387
Title: Streamlining Radioembolization for Cholangiocarcinoma or Metastatic Liver Cancer ≤ 7 cm : Multicenter Prospective Registry Study
Brief Title: Streamlining Radioembolization for CCC and Metastatic Liver Cancer
Acronym: ISTAR-03
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Cheol Kim, Professor, Seoul National University Hospital
Other Study IDs: 2505-094-1640
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Carcinoma (mCRC); Metastatic Liver Cancer; Cholangiocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- streamlining group: radioembolization is performed without MAA scan

SUMMARY:
TARE uses radioactive microspheres (20-60 μm), which are trapped in tumors due to abnormal vasculature, while normal liver sinusoids (≤15 μm) prevent their passage. However, some microspheres may drain into hepatic veins and reach the lungs, risking radiation pneumonitis. Pre-procedural evaluation with angiography and nuclear imaging (MAA scan with SPECT/CT) is required to calculate lung shunt fraction (LSF). TARE is contraindicated if LSF >20%, and may be used with caution if LSF is 10-20%.

Findings associated with high LSF include large tumors, hepatic vein invasion, TIPS, and dysmorphic intratumoral vessels. In contrast, small or medium sized (<7 cm) cholangiocarcinoma or metastatic liver cancers without hepatic vein invasion or dysmorphic vessels show consistently low LSF (<5%). Over 10 years at SNUH, no cases of radiation pneumonitis have been observed in such patients. Therefore, "streamlining TARE" omits pre-procedural nuclear imaging for this group to reduce procedural delays, reserving nuclear imaging for patients who need it most.

SIR-Spheres (SIRTEX) facilitate single-session TARE as they are provided in a bulk vial, unlike TheraSphere which requires advance preparation based on dosimetry.

Protocol Overview :

Procedure: Same-day angiography, cone-beam CT, and TARE using SIR-Spheres.

Dosimetry: Lung shunt fraction is assumed as 5%, estimated lung dose is capped at 10 Gy.

Tumor dose goal: 80~400 Gy (around 250Gy)(single-compartment MIRD), or 300 ~ 1000 Gy (multi-compartment MIRD). minimal tumor dose by partition dosimetry : 100Gy

Software: Simplicit90Y for planning, Y90 PET/CT the next day for post-treatment dosimetry.

Follow-up: 1 year; additional treatments follow institutional guidelines.

This streamlined approach maximizes efficiency while maintaining safety in selected patients.

DETAILED DESCRIPTION:
The radioactive microspheres used in TARE (Transarterial Radioembolization) are very small, approximately 20-60 microns in size. Since the liver sinusoids are less than 15 microns in diameter, the microspheres cannot pass through normal liver parenchyma. However, tumors contain abnormally dilated tumor vasculature, allowing the microspheres to pass through the tumor and potentially drain into the hepatic veins. If a large amount of microspheres reaches the lungs, it can lead to radiation pneumonitis, which may result in death.

Pre-procedural evaluation consists of angiography and nuclear medicine imaging. Angiography determines the number of vessels to be treated and the target area, while nuclear medicine imaging is used to evaluate the lung shunt fraction. Therefore, pre-procedural evaluation is performed first: angiography is conducted, macroaggregated albumin (MAA) is injected into the hepatic artery, and scintigraphy and SPECT/CT are performed to assess lung shunting. If the lung shunt fraction exceeds 20%, TARE is not feasible. If the shunt is between 10-20%, TARE feasibility depends on tumor size. Typically, TARE is performed 1-2 weeks after pre-procedural evaluation.

Findings that suggest a high lung shunt fraction include large tumors, hepatic vein invasion, TIPS (transjugular intrahepatic portosystemic shunt), and dysmorphic intratumoral vessels. Dysmorphic intratumoral vessels are very rare in metastatic liver cancer and intrahepatic cholangiocarcinoma. As both are adenocarcinomas, they typically have lower tumor vascularity compared to hepatocellular carcinoma, resulting in a lower lung shunt fraction. According to Seoul National University Hospital's experience over the past 10 years, mCRC and cholangiocarcinoma less than 7 cm in size, without hepatic vein invasion or dysmorphic intratumoral vessels, almost always showed a lung shunt fraction below 5%. Furthermore, when the tumor is under 7 cm, the treatment area is small, requiring less radiation activity, and the risk of radiation pneumonitis is nearly absent. In the past decade, there have been no cases of radiation pneumonitis in such patients. Therefore, at Seoul National University Hospital, TARE is performed without pre-procedural evaluation in patients meeting the above criteria. This approach is referred to as "streamlining TARE." Recently in Korea, the number of TARE procedures has rapidly increased. To conduct pre-procedural evaluations, scintigraphy and SPECT/CT must be performed by the nuclear medicine department. However, the number of examinations has reached capacity, causing delays in nuclear imaging, which in turn delays TARE procedures in many university hospitals. If TARE is performed without pre-procedural evaluation in patients with small tumors, patients with larger tumors-who truly require evaluation-can undergo it earlier, thus avoiding delays in TARE. Therefore, it is necessary to implement streamlining TARE for metastatic liver cancer or cholangiocarcinoma smaller than 7 cm without dysmorphic intratumoral vessels.

There are two types of radioactive microspheres used in TARE. TheraSphere (Boston Scientific) requires ordering vials with specific radiation activity tailored to each vessel, which necessitates performing pre-procedural evaluation (angiography + nuclear imaging) in advance. On the other hand, SIR-Spheres (SIRTEX) are shipped to hospitals as a mother vial containing more than 7 GBq. The treating hospital determines the number of daughter vials and the necessary radiation activity during the procedure. Therefore, it is possible to perform angiography, determine the number of vessels and required radiation activity, and then proceed with TARE using SIR-Spheres in a single session.

Radioembolization protocol On the day of the procedure, angiography is performed, followed by cone-beam CT of the hepatic artery. The treatment dose is determined using either the single-compartment MIRD or the multi-compartment MIRD method. The lung shunt fraction is assumed to be 5%, and the lung absorbed dose is kept at or below 10 Gy. TN ratio is assumed to be 3.

When using single-compartment MIRD, the mean absorbed dose in the treatment area should range between 80 and 400 Gy, with a target of approximately 250 Gy whenever possible. When using multi-compartment dosimetry, the tumor absorbed dose must be at least 100 Gy and should ideally be within the range of 300 to 600 Gy. While there is no upper limit for the tumor absorbed dose, the lung dose must strictly be kept at or below 10 Gy.

A tumor absorbed dose of ≥300 Gy is defined as boosted TARE, while a dose between 100-300 Gy is defined as regular TARE.

The device used for radioembolization is limited to SIR-Spheres, and the dosimetry is planned using the personalized dosimetry software Simplicit90Y (Mirada).

For treatment beyond the typical scope of radiation segmentectomy, the approach follows the method of Radiation Major Hepatectomy, used for large hepatocellular carcinomas.

Y90 PET/CT is performed on the next day. Post-treatment dosimetry is calculated with Y-90 PET/CT by partition dosimetry.

After radioembolization, patients are followed for one year according to a predefined schedule. During the clinical trial follow-up period, if residual or recurrent tumors are observed, further treatment is administered according to each institution's standard clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 19 and over

  * metastatic liver cancer or cholangiocarcinoma

    * the diameter of the largest tumor ≤ 7cm, tumor number 5 or less

      * FLR volume > 30% of total non-tumorous liver volume

        * Dysmorphic intratumoral vessel : absent, if present, 3mm or thinner ⑥ Child-Pugh class A

          * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 ⑧ No major organ dysfunction according to blood test performed within two months of study enrollment A. Leukocytes ≥ 1,000/µL and ≤ 20,000/µL B. Hemoglobin ≥ 6.0 g/dL (transfusion allowed to meet this criterion) C. Total bilirubin ≤ 2.0 mg/dL D. Platelet ≥ 40,000/µL E. International normalized ratio (INR) ≤ 2.0 for patients not taking anticoagulants F. Aspartate transaminase (AST) ≤ 800 IU/L (i.e., ≤ 20X upper normal limit) G. Alanine transaminase (ALT) ≤ 800 IU/L (i.e., ≤ 20X upper normal limit) H. Creatinine ≤ 2.5 mg/dL (If patients is undergoing hemodialysis, no limit of creatinine) ⑨ Patients with a life expectancy of more than 3 months ⑩ For women of childbearing age, a negative serum pregnancy test. ⑪ Patients who have adequately understood the clinical trial and consented in writing

Exclusion Criteria:

* hepatic vein invasion on dynamic computed tomography (CT) or magnetic resonance imaging (MRI)
* Hepatic vein enhancement on arterial phase CT/MRI
* dysmorphic intratumoral vessel > 3mm on arterial phase CT/MRI
* TIPS is present
* Lobar portal vein enhancement on arterial phase CT/MRI due to AP shunt
* main portal vein tumor thrombosis
* Cases where the operator judges that the occurrence of even mild radiation pneumonitis could be fatal, based on marked emphysema or interstitial lung disease findings on chest CT
* biliary stent or bilioenteric anastomosis
* History of severe allergy of intolerance to contrast agents
* Contraindication to angiography or selective visceral catheterization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic liver cancer or cholangiocarcinoma who are scheduled for radioembolization
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-22 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate according to the localized RECIST criteria | up to 1 year

SECONDARY OUTCOMES:
Overall survival (OS) rates | From date of radioembolization until the date of death from any cause, assessed up to 60 months
Progression free survival (PFS) rates according to RECIST and localized RECIST | From date of radioembolization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
AE and serious adverse event (SAE) according to CTCAE v5.0 | Time of treatment up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
The presence or absence of radiation pneumonitis diagnosed by chest simple X-ray or CT | Time frame: Time of treatment up to 180 days after the initial treatment or subsequent anticancer treatment, whichever comes first

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance hospital, Seoul

IPD SHARING:
Plan to Share IPD: No